CLINICAL TRIAL: NCT06601413
Title: Modified Thoracoabdominal Nerves Block Through Perichondrial Approach (M-TAPA) Versus Incisional Local Anesthetic Administration for Total Laparoscopic Hysterectomy : a Prospective, Randomized Clinical Study
Brief Title: Modified Thoracoabdominal Nerve Block(M-TAPA) in Total Laparoscopic Hysterectomies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ELA ERTEN, medical doctor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-KAEK-159
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain,Postoperative
Keywords: M-TAPA, post-operative pain,; Total laparoscopyc histerectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M-TAPA Group (Active Comparator): At the end of the surgery, without waking the patient, a linear transducer will be placed on the costochondral angle in the sagittal plane under ultrasound guidance, and a total of 40 mL of LA (0.25% Bupivacaine) will be applied bilaterally to the lower surface of the chondrium, giving a deep angle to see the lower side of the chondrium centrally.
  Interventions: Other: M-TAPA Block
- Trochar-site Group (Placebo Comparator): At the end of surgery, infiltration analgesia will be applied by the surgeon to all trocar entry sites (4 port entries) with 10 ml of 0.25% bupivacaine (40 mL in total) without waking the patient.
  Interventions: Other: Trocar site local anesthetic infiltration

INTERVENTIONS:
Other: M-TAPA Block — M-TAPA block will administer ultrasound guided (Sonosite, Inc., Bothell, WA, USA) bilaterally by same anesthesiologist (E.E.) who had more than 10 years experience of regional anesthesia, before weaking from general anesthesia after the surgical procedure. A high-frequency (6-13 MHz) linear probe (HFL38) will be used to identify the transversus abdominis, internal oblique, and external oblique muscles on the costochondral angle in the sagittal plane at the 10th costal margin. In the midclavicular line, between the upper fascia of the transversus abdominis muscle and the lower fascia of the costochondral tissue, at the level of the 10th rib, 20 mL of 0.25 percent bupivacaine will be injected (arcus costarum). The same procedure will be followed on the other side.
  Arms: M-TAPA Group
Other: Trocar site local anesthetic infiltration — At the end of surgery, infiltration analgesia will be applied to all trocar entry sites (4 port entries) by the surgeon with 10 ml of 0.25% bupivacaine (40 mL in total) without waking the patient.
  Arms: Trochar-site Group

SUMMARY:
The aim of the study is comparing the postoperative effects of ultrasound-guided Modified Perichondrial Approach to Thoracoabdominal Nerves (M-TAPA) block for postoperative pain control after total laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Pain is one of the most common problems seen in the postoperative period in patients who underwent total laparoscopic hysterectomy.

Multimodal analgesia methods are used in postoperative pain management. Nerve blocks, which are an important component of multimodal analgesia, have an important place in postoperative analgesia management today.

Local Anesthetic Infiltration at the Trocar Site is the most classical nerve block method that has been used for a long time as a part of multimodal analgesia in laparoscopic surgeries.

Modified TAPA block applied with ultrasound guidance; It is a regional block affecting both the anterior and lateral branches of the thoracoabdominal nerves with a perichondrial approach. It is used in total laparoscopic hysterectomies.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Elective cases
* ASA I-III functional status
* Body mass index (BMI)<35
* Total laparoscopic hysterectomy planned with general anesthesia
* No contraindications for M-TAPA block to be applied
* Cases that give written and verbal consent for participation in the study will be included.

Exclusion Criteria:

* Conversion to open surgery
* Development of perioperative complications (due to surgery and/or anesthesia)
* Coagulation disorder
* Infection at the injection site
* Allergy to local anesthesia
* Those who used any painkillers in the preoperative 24 hours
* Those who did not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 66 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative total tramadol consumption for first 24 hours | Postoperative 24 hours
  The intravenous PCA pump will be programmed to deliver a bolus of 20 mg tramadol with a lockout interval of 30 min and no baseline infusion (tramadol 500 mg in 100 mL SF

SECONDARY OUTCOMES:
Postoperative pain scores | at postoperative 0 (PACU), 1, 2, 4, 8, 12 and 24 hours
  Pain will be assessed with visual analog score (VAS) in 2 different ways, at rest and with movement (VAS: 0, no pain; 10, worst pain imaginable). VAS scores will be recorded at postoperative 0 (PACU), 1, 2, 4, 8, 12 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No